CLINICAL TRIAL: NCT00007293
Title: Phototherapy of Psoriasis of the Scalp With a UV-B Emitting Fiber Optic Comb
Brief Title: Scalp Psoriasis Treatment With a Fiber Optic Comb
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R44AR044449 (NIH); NIAMS-049
Record Dates: First submitted 2000-12-16; First posted 2000-12-18 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2003-02

CONDITIONS: Psoriasis
Keywords: Phototherapy; Psoriasis; Scalp psoriasis; Fiber optic; Light comb; UV source
MeSH Terms: conditions — Psoriasis

INTERVENTIONS:
Device: UV-B Lightsource and Fiber Optic Comb

SUMMARY:
This study will test the safety and effectiveness of a novel fiber optic device for treating scalp psoriasis with ultraviolet (UV-B) light. A effective treatment is not currently available for people with scalp psoriasis. Present methods for treating psoriasis with UV-B light cannot be used for the scalp because hair is usually blocking the light from reaching the affected skin. Our method overcomes this problem with the use of a comb that has optical fibers to deliver light directly to the skin. We will evaluate this device in a clinical setting and will use the results to tailor the design of the comb before producing it in large quantities.

DETAILED DESCRIPTION:
Scalp psoriasis can be treated with a novel fiber optic delivery system that irradiates the psoriatic scalp of patients with UV-B light via an optical fiber comb. Current methods for treatment of psoriasis with light are not applicable to the scalp because hair is usually blocking the light from reaching the affected skin. Our method overcomes this problem with the use of a comb that has optical fibers to deliver light directly to the skin. We have developed a UV-B light source and a fiber optic comb for use in clinics and doctors' offices. We will evaluate this device in a clinical setting.

The results of this trial will provide data about the effectiveness of the device. We will use these results to tailor the design before it is ready for volume production. If successful, the UV-B light source and fiber optic comb will provide treatment to people affected with scalp psoriasis. At present, these people do not have any effective treatment available to them.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either sex and any race or ethnic background with chronic, stable, bilateral psoriasis of the scalp.

Exclusion Criteria:

* Subjects who are currently taking systemic medications for psoriasis (e.g., methotrexate, retinoids).
* Subjects who are currently using or have used topical medications other than emollients in the past 6 weeks on their scalp.
* Patients with pustular psoriasis, known photosensitivity disorders, lupus erythematosus, or unstable major illnesses preventing participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2000-08; Study Completion 2002-07

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Taneja A, Racette A, Gourgouliatos Z, Taylor CR. Broad-band UVB fiber-optic comb for the treatment of scalp psoriasis: a pilot study. Int J Dermatol. 2004 Jun;43(6):462-7. doi: 10.1111/j.1365-4632.2004.01993.x. PMID 15186234